CLINICAL TRIAL: NCT02442310
Title: Single Dose Crossover Comparative Bioavailability Study of Deferiprone 600 mg Delayed Release Tablets Versus Deferiprone Oral Solution in Healthy Male and Female Volunteers Following a 1200 mg Dose
Brief Title: Comparison of Deferiprone Delayed Release Tablets and Deferiprone Oral Solution in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ApoPharma (Industry)
Collaborators: Algorithme Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: LA46-0114
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: deferiprone; deferiprone delayed release formulation; pharmacokinetics
MeSH Terms: interventions — Deferiprone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Delayed release, fed conditions (Experimental): A single 1200 mg dose of deferiprone delayed release tablet formulation administered following a high-fat breakfast
  Interventions: Drug: Deferiprone delayed release tablet formulation
- Delayed release, fasting conditions (Experimental): A single 1200 mg dose of deferiprone delayed release tablet formulation, administered following a 10-hour fast
  Interventions: Drug: Deferiprone delayed release tablet formulation
- Delayed release half-tablets (Experimental): A single 1200 mg dose of deferiprone delayed release tablet formulation, following a high-fat breakfast
  Interventions: Drug: Deferiprone delayed release tablet formulation
- Oral solution, fasting conditions (Active Comparator): A single 1200 mg dose of deferiprone oral solution, administered following a 10-hour fast
  Interventions: Drug: Deferiprone oral solution

INTERVENTIONS:
Drug: Deferiprone delayed release tablet formulation — Deferiprone 600 mg delayed release tablet formulation
  Other Names: Deferiprone
  Arms: Delayed release half-tablets; Delayed release, fasting conditions; Delayed release, fed conditions
Drug: Deferiprone oral solution — Deferiprone 100 mg/mL oral solution
  Other Names: Ferriprox
  Arms: Oral solution, fasting conditions

SUMMARY:
The purpose of this study is to look at the pharmacokinetics of a new formulation of deferiprone (deferiprone delayed release tablets) under fed and fasting conditions.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, 4-period crossover study of the pharmacokinetics of a new formulation of deferiprone, delayed release tablets in twenty healthy volunteers. In each study period, blood samples for pharmacokinetics assessment will be collected pre-dose and over 24 hours post-dose. Safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 to <50 years
2. A female volunteer of childbearing potential must agree to use an accepted contraceptive regimen from at least 28 days prior to the first administration of the study drug until at least 30 days after the last dose of the study drug
3. A sexually active male must agree that he and/or his female partner will use a medically acceptable method of contraception throughout the study and for at least 30 days following drug administration
4. Body mass index (BMI) greater than or equal to 18.5 kg/m^2 and below 30.0 kg/m^2
5. Non- or ex smoker
6. Clinical laboratory values within the laboratory's stated normal range; if not within this range, an abnormal value must be without any clinical significance
7. Have no clinically significant diseases captured in the medical history, or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, general biochemistry, coagulation, ECG, and urinalysis)

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Absolute neutrophil count (ANC) < 1.8 x 109/L at screening (no repeat can be performed)
3. History of significant hypersensitivity to deferiprone or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (such as angioedema) to any drugs
4. History or presence of gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
5. Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
6. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 220 msec, QRS < 60 msec, QRS >119 msec and QTcF > 450 msec for males and > 460 msec for females) on the screening ECG or other clinically significant ECG abnormalities
7. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
8. Any clinically significant illness in the previous 28 days before Day 1 of this study
9. Serum ferritin value below the normal limit of the reference laboratory at screening
10. Positive urine screening of alcohol and/or drugs of abuse
11. Positive results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG (B) (hepatitis B)) or anti-Hepatitis C Virus (HCV (C)) tests

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Tricta, MD, Study Chair — ApoPharma Inc.
Locations (1):
- Algorithme Pharma Inc., Mount Royal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: Subjects were randomized to receive the following four treatments in different orders, with a 7-day washout period between treatments:
  * Deferiprone delayed release tablets under fed conditions.
  * Deferiprone delayed release tablets under fasting conditions.
  * Deferiprone delayed release tablets administered as half-tablets, under fed conditions.
  * Deferiprone oral solution under fasting conditions
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 20
Completed | 17
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Region of Enrollment [Number; unit: participants]
  Canada | 20

OUTCOME MEASURES:

1. Primary Outcome: Cmax for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Maximum measured serum concentration. Blood samples will be collected pre-dose and over a 24-hour interval post-dose
Time Frame: 24-hour interval
Population: The pharmacokinetics population included all subjects who provided evaluable data for at least one of the comparisons of interest
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Delayed Release, Fed Conditions | Delayed Release, Fasting Conditions | Delayed Release Half-tablets | Oral Solution, Fasting Conditions
Number analyzed (Participants) | 18 | 17 | 18 | 17
μg/mL
  Cmax for serum deferiprone | 8.05 (2.85) | 8.21 (2.18) | 7.43 (2.00) | 16.71 (4.54)
  Cmax for serum deferiprone 3-O-glucuronide | 15.77 (3.80) | 19.27 (3.73) | 15.40 (4.33) | 21.87 (4.34)

2. Primary Outcome: Tmax for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Time to maximum observed serum concentration. Blood samples will be collected pre-dose and over a 24-hour interval post-dose
Time Frame: 24-hour interval
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Delayed Release, Fed Conditions | Delayed Release, Fasting Conditions | Delayed Release Half-tablets | Oral Solution, Fasting Conditions
Number analyzed (Participants) | 18 | 17 | 18 | 17
Hour
  Tmax for serum deferiprone | 3.93 (1.77) | 2.05 (0.60) | 3.49 (1.68) | 0.52 (0.16)
  Tmax for serum deferiprone 3-O-glucuronide | 4.63 (1.48) | 3.03 (0.52) | 4.75 (1.87) | 1.87 (0.34)

3. Primary Outcome: AUC0-∞for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Area under the serum concentration time curve extrapolated to infinity. Blood samples will be collected pre-dose and over a 24-hour interval post-dose
Time Frame: 24-hour interval
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Delayed Release, Fed Conditions | Delayed Release, Fasting Conditions | Delayed Release Half-tablets | Oral Solution, Fasting Conditions
Number analyzed (Participants) | 17 | 17 | 17 | 17
ug*h/mL
  AUC0-∞ for serum deferiprone | 36.70 (9.37) | 35.77 (8.74) | 37.18 (9.72) | 40.61 (10.72)
  AUC0-∞ for serum deferiprone 3-O-glucuronide | 97.52 (11.47) | 100.44 (13.49) | 98.23 (10.64) | 101.34 (13.99)

4. Secondary Outcome: Number of Subjects With Adverse Events (AEs)
Description: Number of subjects with AEs, by frequency, severity, time to onset, duration, and relatedness to study product. AEs will include clinically significant changes from baseline in vital signs, 12-lead ECG, physical examinations, and laboratory tests.
Time Frame: Throughout the trial, from the time of the first dose until the last study visit (Day 30 or early termination)
Population: The safety population included all subjects who received at least one of the investigational products under study.
Measure: Number; unit: participants
Arm/Group | Delayed Release, Fed Conditions | Delayed Release, Fasting Conditions | Delayed Release Half-tablets | Oral Solution, Fasting Conditions
Number analyzed (Participants) | 18 | 18 | 19 | 17
participants | 3 | 4 | 5 | 6

ADVERSE EVENTS:
Arm/Group | Delayed Release, Fed Conditions | Delayed Release, Fasting Conditions | Delayed Release Half-tablets | Oral Solution, Fasting Conditions
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 3/18 | 4/18 | 5/19 | 6/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Release, Fed Conditions (N=18) | Delayed Release, Fasting Conditions (N=18) | Delayed Release Half-tablets (N=19) | Oral Solution, Fasting Conditions (N=17)
Vessel Puncture Site Haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Face Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel Puncture Site Bruise (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Amylase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paresthesia Mucosal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor retained title to and the right to publish all documentation, records, raw data, specimens or other work product generated in connection with the trial. Such publications shall not be made without the prior written consent of Sponsor. Neither Party will use the other Party's name in connection with any publication or promotion without the other Party's prior written consent. However, Sponsor has the right to publish appropriate information in order to satisfy regulatory requirements.